CLINICAL TRIAL: NCT03925909
Title: Effect of Chronic Eriocitrin Supplementation on the Intestinal Microbiota of Pre-diabetic and Insulin Resistant Individuals
Brief Title: Supplementation of Eriocitrin in Intestinal Microbiota
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because there was no funding
Sponsor: São Paulo State University (Other)
Responsible Party: Principal Investigator, Thais Cesar, Principal Investigator, São Paulo State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SaoPSU 13
Record Dates: First submitted 2019-04-17; First posted 2019-04-24 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Pre Diabetes
Keywords: Eriocitrin; Citrus bioflavonoids; Flavanone; Pre-diabetes; Blood glucose; Microbiome
MeSH Terms: conditions — Glucose Intolerance | interventions — eriocitrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Eriomin 200 mg (Experimental): The volunteers will receive one capsule containing 200 mg eriocitrin
  Interventions: Dietary Supplement: Eriocitrin
- Eriomin 400 mg (Experimental): The volunteers will receive one capsule containing 400 mg eriocitrin
  Interventions: Dietary Supplement: Eriocitrin
- Eriomin 800 mg (Experimental): The volunteers will receive one capsule containing 800 mg eriocitrin
  Interventions: Dietary Supplement: Eriocitrin
- Placebo (No Intervention): The volunteers will receive a capsule containing corn starch (placebo)

INTERVENTIONS:
Dietary Supplement: Eriocitrin — The responsible nutritionists will do 1) Anthropometric Assessment, in which weight data will be collected (kg); height (m); waist circumference (cm), waist circumference (cm) and hip circumference (cm), muscle mass (kg /%) and percentage of fat by means of bioimpedance equipment; 2) Dietary assessment, which will be performed through a 24-hour Food Recall, a 3-day Food Record and a Food Consumption Frequency Questionnaire; 3) Evaluation of the microbiota, for which stool will be collected from the last 24 hours on the day before the beginning of the experiment and at the end of the study (week 12); 3) Biochemical evaluation, which includes the collection of 30 mL of blood to be performed by trained and qualified technicians.
  Arms: Eriomin 200 mg; Eriomin 400 mg; Eriomin 800 mg

SUMMARY:
Pre-diabetes is characterized by high plasma concentration of glucose and glycated hemoglobin and is the main risk factor for the development of type 2 diabetes. Several studies show that the intestinal microbiota is intimately linked to cardio-metabolic factors (type 2 diabetes, insulin resistance) when in situations of dysbiosis. Food is a key element for a healthy microbiota, focusing on the consumption of polyphenols that modulate the intestinal environment through its alteration and production of short chain fatty acids, and can thus be a way of reversing situations such as pre- diabetes and insulin resistance. The objective of the study will be to investigate whether chronic supplementation of eriocitrin alters the intestinal microbiota of pre-diabetic and insulin resistant individuals, reversing these situations. This will be done by supplementation of eriocitrin-containing capsules with different dosages in pre-diabetic and insulin resistant individuals. There will be 12 weeks of intervention, with faecal collections, anthropometric and dietary evaluation, and then will be made microbiological analysis to identify the intestinal microbiota and biochemical analysis before and after the intervention. For statistical analysis, normality and homogeneity test (Kolmogorov-Smirnov and Levine test respectively), T-test to compare baseline time between groups and repeated-measures ANOVA (two-way) were used to compare changes within and between groups.

DETAILED DESCRIPTION:
Individuals of both sexes between 30 and 60 years of age who present fasting glycemia between 100 mg / dL (5,6 mmol / L) and 125 mg / dL (6,9 mmol / L) 50, or concentration of glycated hemoglobin between 5.7% (39 mmol / mole) and 6.4% (47 mmol / mole) 50, or glycemic concentrations in the oral glucose tolerance test between 140mg / dL (7.8 mmol / L) to 199mg / dL (11.0 mmol / L) 50. The study will also include insulin-resistant individuals: insulin above 25 uU / mL, or who present HOMA-IR score above 2.7.

Individuals using supplements (vitamins, bioflavonoids), pregnant women and those who practice intense physical exercise (> 10h / week) will be excluded from the study.

The primary endpoint will be alteration of the microbiota with possible improvement of the glycemic profile, leading to the reversal of pre-diabetes and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* 30-60 years
* Increased fasting blood glucose from 6.1 to 7.0 mmol / L or,
* Decreased glucose tolerance of 7 , 8 to 11.1 mmol / L or,
* Glycated hemoglobin with values between 5.7 and 6.4%

Exclusion Criteria:

* Use hypoglycemic, hypolipidemic drugs,
* Use dietary supplements (vitamins, minerals, bioflavonoids, prebiotics, probiotics or other bioactive compounds),
* Exercise intensely (more than 10 hours per week)
* History of cardiovascular diseases , diabetes mellitus, liver and kidney disease.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Rate of change in microbiome | 0-12 week
  Changes in microbiome before and after administration of the intervention / placebo

SECONDARY OUTCOMES:
Rate of change in plasma glucose concentration | 0-12 week
  Changes in serum 2 hours after oral glucose tolerance test, HbA1c, insulin, HOMA-IR before and after administration of the intervention / placebo

CONTACTS AND LOCATIONS:
Overall Officials: Thais B Cesar, Phd, Principal Investigator — ao Paulo State University "Julio de Mesquita Filho"
Locations (1):
- Sao Paulo State University "Julio de Mesquita Filho", Araraquara, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No